CLINICAL TRIAL: NCT03345108
Title: A Randomized, Open-Label, Clinical Study to Evaluate a Methodology to Assess Food Occlusion Efficacy of a Denture Adhesive in Healthy, Edentulous Subjects
Brief Title: A Study to Investigate a Method to Measure Food Occlusion by Denture Adhesives in Denture Wearers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 208397
Record Dates: First submitted 2017-11-13; First posted 2017-11-17 (Actual); Results first posted 2019-03-29 (Actual); Last update posted 2019-03-29 (Actual); Status verified 2019-03

CONDITIONS: Denture Retention

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Test Denture Adhesive (Conventional Application) (Experimental): Test denture adhesive will be applied to participants' dentures via conventional pattern of application.
  Interventions: Device: Denture Adhesive Cream (Conventional Application)
- Test Denture Adhesive (Continuous strip Application) (Experimental): Test denture adhesive will be applied to participants' dentures via continuous strips pattern of application.
  Interventions: Device: Denture Adhesive (Continuous Strip Application)
- Negative Control (Other): Participants will not apply any denture adhesive in this treatment arm.
  Interventions: Other: No Adhesive

INTERVENTIONS:
Device: Denture Adhesive Cream (Conventional Application) — The adhesive cream will be extruded from a pre-dosed syringe. 1.6 g of adhesive per treatment will be applied to each participant's dentures. This dose will be split as 1.00±0.05g for the maxillary and 0.60±0.05g for the mandibular dentures.
  Arms: Test Denture Adhesive (Conventional Application)
Device: Denture Adhesive (Continuous Strip Application) — The adhesive cream will be extruded from a pre-dosed syringe. 1.6 g of adhesive per treatment will be applied to each participant's dentures. This dose will be split as 1.00±0.05 g for the maxillary and 0.60±0.05 g for the mandibular dentures.
  Arms: Test Denture Adhesive (Continuous strip Application)
Other: No Adhesive — No adhesive applied.
  Arms: Negative Control

SUMMARY:
The purpose of this study is to evaluate a methodology to determine the ability of a denture adhesive to restrict food ingress underneath dentures during eating.

DETAILED DESCRIPTION:
This will be a single centre, controlled, open label, randomized, three-treatment, three-period, cross-over design in participants with full upper and full lower dentures. Each treatment period will consist of one day of testing with at least two days between adjacent treatment visits. This study will consist of four visits: Visit 1 - Screening Visit; Visit 2 - Treatment 1 Visit; Visit 3 - Treatment 2 Visit and Visit 4 - Treatment 3 Visit. (Participants will use Test product (denture adhesive) applied to the dentures either in a pattern consistent with standard application or applied to the dentures in a pattern of continuous strips. Participants will also use no adhesive as a control. Participants will cross-over between treatments so that all participants will participate in all 3 treatment arms. An hour after the participant has worn their denture, they will chew a portion of peanuts in a controlled manner. The peanuts that migrate under the denture during this chewing procedure will be collected, washed, dried and weighed. Participant will also answer a short questionnaire on the procedure and record the number of times their denture dislodged during the chewing procedure. The study hypothesis is that this methodology will enable comparisons between denture adhesives and no adhesive to demonstrate the effectiveness of denture adhesives at restricting food ingress under dentures during eating.

ELIGIBILITY:
Inclusion Criteria:

* Evidence of a personally signed and dated informed consent document indicating that the participant has been informed of all pertinent aspects of the study before any assessment is performed.
* Male or female who, at the time of screening, are between the ages of 18 and 85 years, inclusive.
* Willing and able to comply with scheduled visits, treatment plan, and other study procedures.
* Healthy, defined as in general good physical health, as judged by the investigator.
* Self-reports experience of getting food trapped under their denture.
* Is an habitual wearer of both of their dentures defined as participants who wear both of their dentures for the majority of their time whilst awake.
* Females of childbearing potential and at risk for pregnancy must agree to use a highly effective method of contraception throughout the study and for 1 day after the last dose of assigned treatment.
* Female participants who are not of childbearing potential must meet following requirements: a) Achieved postmenopausal status, defined as follows: cessation of regular menses for at least 12 consecutive months with no alternative pathological or physiological cause; status may be confirmed by having a serum follicle stimulating hormone (FSH) level confirming the post-menopausal state, b) Have undergone a documented hysterectomy and/or bilateral oophorectomy, and have medically confirmed ovarian failure.
* Have denture prostheses that fulfil all of the following: a) A qualifying conventional acrylic full denture in both the upper and lower arch, b) Dentures are well fitting (Kapur (Olshan Modification) Retention and Stability Index Sum Score ≥6) (Olshan, 1992) with no individual stability or retention scores <1, c) Dentures are well made (according to the well-made assessment), and d) Has a peanut particle migration rating >0 for each denture.

Exclusion Criteria:

* An investigational site staff member directly involved in the conduct of the study or their family member, site staff members otherwise supervised by the investigator, or an employee of the sponsor directly involved in the conduct of the study.
* Participation in any other clinical study involving investigational drugs, cosmetics or medical devices within 30 days prior to study entry and/or during study participation.
* Acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the participant inappropriate for entry into this study.
* Pregnant female participants.
* Breastfeeding female participants.
* Known or suspected intolerance or hypersensitivity to the study materials (or closely related compounds) or any of their stated ingredients.
* Unwilling or unable to comply with the Lifestyle Guidelines described in this protocol.
* History of swallowing difficulties or choking.
* Currently taking or have taken a bisphosphonate drug (i.e., Fosamax®, Actonel®, Boniva®) for treatment of osteoporosis.
* Any clinically significant or relevant oral abnormality (e.g. temporomandibular joint [TMJ] problems) that, in the opinion of the investigator, could affect the participants participation in the study.
* Known allergy to peanuts or any other nut.
* Any condition or medication which, in the opinion of the investigator, is currently causing xerostomia.
* Recent history (within the last year) of alcohol or other substance abuse.
* OST examination findings such as stomatitis, open sores, lesions, redness or swelling which in the opinion of the investigator, would interfere with the conduct of the study.
* Use of any medication that, in the opinion of the investigator, would interfere with the conduct of the study.
* A serious chronic disease requiring intermittent hospital visits.
* Having been previously enrolled in this study.
* Any participant who, in the opinion of the investigator, should not participate in the study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2017-11-20 (Actual); Primary Completion 2017-12-15 (Actual); Study Completion 2017-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline; GSK Clinical Trials, Study Director — GlaxoSmithKline (for GlaxoSmithKline; Human Genome Sciences Inc., a GSK Company; Sirtris, a GSK Company; Stiefel, a GSK Company; ViiV Healthcare)
Locations (1):
- GSK Investigational Site, Fort Wayne, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All the participants were recruited from one center in United States.
Pre-assignment Details: A total of 49 participants were screened for entry into the study, of whom 48 were randomized. 1 participant did not meet the study criteria. Out of 48, only 47 subjects started the no adhesive treatment period, since 1 participant discontinued the study due a scheduling (withdrawal of consent).
Groups:
- A-B-C: Sequence of the treatment if A-B-C, where A-conventional application; B- continuous strip application; C- no adhesive
- A-C-B: Sequence of the treatment if A-C-B, where A-conventional application; B- continuous strip application; C- no adhesive
- B-A-C: Sequence of the treatment if B-A-C, where A-conventional application; B- continuous strip application; C- no adhesive
- B-C-A: Sequence of the treatment if B-C-A, where A-conventional application; B- continuous strip application; C- no adhesive
- C-A-B: Sequence of the treatment if C-A-B, where A-conventional application; B- continuous strip application; C- no adhesive
- C-B-A: Sequence of the treatment if C-B-A, where A-conventional application; B- continuous strip application; C- no adhesive
Period: Period-1
Arm/Group | A-B-C | A-C-B | B-A-C | B-C-A | C-A-B | C-B-A
Started | 8 | 8 | 8 | 8 | 8 | 8
Completed | 8 | 8 | 8 | 8 | 8 | 8
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Period-2
Arm/Group | A-B-C | A-C-B | B-A-C | B-C-A | C-A-B | C-B-A
Started | 8 | 8 | 8 | 8 | 8 | 8
Completed | 8 | 8 | 8 | 8 | 8 | 8
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Period-3
Arm/Group | A-B-C | A-C-B | B-A-C | B-C-A | C-A-B | C-B-A
Started | 7 | 8 | 8 | 8 | 8 | 8
Completed | 7 | 8 | 8 | 8 | 8 | 8
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: 47 participants started the no adhesive treatment period, since 1 participant discontinued the study after completing period 2 and therefore did not return for treatment period 3 of no adhesive. The demographic and baseline characteristics has been reported for intent-to-treat (ITT) population (N=48).
Groups:
- Overall: Includes participants with conventional application of adhesive, continuous strip application of adhesive and no adhesive
Arm/Group | Overall
Number analyzed (Participants) | 48
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.0 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34
  Male | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 44
  More than one race | 0
  Unknown or Not Reported | 0
Current Lower Denture Age [Mean (Standard Deviation); unit: Years] | 11.4 (12.31)
Current Upper Denture Age [Mean (Standard Deviation); unit: Years] | 12.0 (12.25)

OUTCOME MEASURES:

1. Primary Outcome: Mass of Peanuts Under Combined Maxillary and Mandibular Dentures (Denture Adhesive Applied Per Conventional Pattern)
Description: Participants received 1.6 grams (g) of test adhesive on their dentures in a conventional pattern. After 60 minutes (min), participants were provided with 30-32 g non-salted peanuts, divided into smaller portions of approximately eight peanut halves. Each portion chewed for approximately 20 seconds (s). After consumption of all peanuts, participants had rinse their mouth with water for approximately 5 s. Dentures were removed and any peanuts remaining in the mouth were collected using a gauze. Both denture and gauze were placed in a beaker with hot de-ionized water and sonicated for 30 minutes (min) after which the water was strained through a standard testing sieve. The collected particles were washed and air-dried and transferred to pre-weighed aluminium weighing pans using a spatula and then, were dried in an oven at 40-degree Celsius for 5 hours. The pans were removed, cooled to room temperature and then weighed to determine the mass of the particles collected from each denture.
Time Frame: Upto 9 weeks
Population: The primary endpoint has been measured for intent-to-treat (ITT) population (N=48). The ITT population included all randomized participants who received at least 1 dose of study treatment during the study and consumed peanuts and had at least 1 mass of peanuts from both upper and lower dentures.
Measure: Mean (Standard Deviation); unit: Grams
Groups:
- Conventional Application: Participants received the 1.6 grams (g) of adhesive to the denture which was placed in the mouth as 1.0 g for maxillary denture and 0.6 g for mandibular denture. In this group, the test denture adhesive was applied in conventional pattern which is defined as the adhesive was filled in pre-weighed syringe and was applied in short strips (3 strips to the upper denture and 2 strips on the lower denture), not too close to the denture. Participants rinsed their mouth before inserting the dentures and bit down for few seconds to secure hold.
- Continuous Strip Application: Participants received the 1.6 g of adhesive to the denture which was placed in the mouth as 1.0 g for maxillary denture and 0.6 g for mandibular denture. In this group, the test denture adhesive was applied in continuous strip pattern which is defined as the adhesive was filled in pre-weighed syringe and was applied in long, continuous strips (3 strips to the upper denture and 1 strip on the lower denture), not too close to the denture. Participants rinsed their mouth before inserting the dentures and bit down for few seconds to secure hold.
- No Adhesive: Participants did not receive any denture adhesive in this group.
Arm/Group | Conventional Application | Continuous Strip Application | No Adhesive
Number analyzed (Participants) | 48 | 48 | 47
Grams | 0.01184 (0.016237) | 0.00944 (0.013326) | 0.07853 (0.158567)

ADVERSE EVENTS:
Time Frame: 95 days
Arm/Group | Conventional Application | Continuous Strip Application | No Adhesive
All-Cause Mortality (participants affected / at risk) | 0/48 | 0/48 | 0/47
Serious Adverse Events (participants affected / at risk) | 0/48 | 0/48 | 0/47
Other Adverse Events (participants affected / at risk) | 0/48 | 0/48 | 0/47

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-10-24): https://cdn.clinicaltrials.gov/large-docs/08/NCT03345108/Prot_000.pdf
  • Statistical Analysis Plan (2017-12-14): https://cdn.clinicaltrials.gov/large-docs/08/NCT03345108/SAP_001.pdf